CLINICAL TRIAL: NCT04730895
Title: Investigating the Role of 13cis Retinoic Acid in the Treatment of COVID-19 and Enhancement of Its Spike Protein Based Vaccine Efficacy and Safety.
Acronym: Isotretinoin
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Faculty of Science, Damietta University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COVID vaccine
Record Dates: First submitted 2021-01-28; First posted 2021-01-29 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Covid19 Vaccine
MeSH Terms: interventions — Isotretinoin; ChAdOx1 nCoV-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Oral 13 cis retinoic acid (Experimental): The participants will receive 13 cis retinoic acid (0.5 mg/kg/day in 2 divided doses orally for 14 days . All subjects were encouraged to complete the full course of treatment and common side effects were explained. Side effects and compliance will be documented.
  Interventions: Drug: Oral 13 cis retinoic acid
- Aerosolized 13 cis retinoic acid (Experimental): The participants will receive Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days. All subjects were encouraged to complete the full course of treatment and common side effects were explained. Side effects and compliance will be documented.
  Interventions: Drug: Aerosolized 13 cis retinoic acid
- 13 cis retinoic acid doses orally in combination with spike protein based vaccine (Experimental): The participants will receive 13 cis retinoic acid (0.5 mg/kg/day in 2 divided doses orally for 14 days and also, participants will receive two doses of spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine in deltoid of non-dominant arm, 28 days apart. Participants will have 15 routine visits over a 24 month period.All subjects were encouraged to complete the full course of treatment and common side effects were explained. Side effects and compliance will be documented
  Interventions: Combination Product: 13 cis retinoic acid doses orally in combination with spike protein based vaccine
- Aerosolized 13 cis retinoic acid in combination with spike protein based vaccine (Experimental): The participants will receive Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days and also, participants will receive two doses of 5-7.5x10^10 vp spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine in deltoid of non-dominant arm, 28 days apart. Participants will have 15 routine visits over a 24 month period.All subjects were encouraged to complete the full course of treatment and common side effects were explained. Side effects and compliance will be documented
  Interventions: Combination Product: Aerosolized 13 cis retinoic acid in combination with spike protein based vaccine
- spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine (Sham Comparator): The participants will receive two doses of 5-7.5x10^10 vp spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine in deltoid of non-dominant arm, 28 days apart. Participants will have 15 routine visits over a 24 month period.All subjects were encouraged to complete the full course of treatment and common side effects were explained. Side effects and compliance will be documented
  Interventions: Biological: Biological: spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine

INTERVENTIONS:
Drug: Oral 13 cis retinoic acid — Dose of 0.5 mg/kg/day in 2 divided doses orally for 14 days
  Arms: Oral 13 cis retinoic acid
Drug: Aerosolized 13 cis retinoic acid — Dose of Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases froms 0.2 mg/kg/day to 4 mg/kg/day
  Arms: Aerosolized 13 cis retinoic acid
Combination Product: 13 cis retinoic acid doses orally in combination with spike protein based vaccine — Dose of 13 cis retinoic acid (0.5 mg/kg/day in 2 divided doses orally for 14 days and also, participants will receive two doses of 5-7.5x10^10 vp spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine in deltoid of non-dominant arm, 28 days apart
  Arms: 13 cis retinoic acid doses orally in combination with spike protein based vaccine
Combination Product: Aerosolized 13 cis retinoic acid in combination with spike protein based vaccine — Dose of Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day for 14 days and also, participants will receive two doses of 5-7.5x10^10 vp spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine in deltoid of non-dominant arm, 28 days apart
  Arms: Aerosolized 13 cis retinoic acid in combination with spike protein based vaccine
Biological: Biological: spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine — Dose of 5-7.5x10^10vp of spike protein based vaccine such as ChAdOx1 nCoV-19 in deltoid of non-dominant arm, 28 days apart
  Arms: spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine

SUMMARY:
Investigating the role of 13cis retinoic acid in the treatment of COVID-19 and enhancement of Its spike protein based vaccine efficacy and safety.

DETAILED DESCRIPTION:
The study is an urgent randomized interventional comparative Phase II trial for investigating the expected long term side effects of spike protein based vaccine which may vary from thrombosis, platelet aggregation, autoantibodies against ACE2, to lung damage and other ACE2 expressing cell damage. This clinical study is conducted on 360 adult male and female participants, Here, we submitted this clinical trial depending on studies with up to date literature guidance to indicate that 13 cis Retinoic Acid will provide complete protection against COVID-19 and will be better option for effective and safe COVID-19 vaccine owing to its ability to induce mucosal IgA antibodies that are less prone to ADE phenomenon and responsible for passive mucosal immunity in the respiratory tract. Retinoic acid strengthens mucosal immunity via inducing IgA antibodies and considered potent IgA isotype Furthermore, its impact on ACE2 receptors, Memory T cells, CD4+/CD8+ ratio, Neutrophil Chetnotaxis, Interferon Type1, Thrombin, Transmembrane serine protease 2 (TMPRSS2), toll-like receptor 3 (TLR3), mitochondrial antiviral-signaling protein (MAVS), papain-like protease (PLpro), and Interleukin 6 ( Il-6).

-----------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------

The SARS-CoV-2 spike protein directly binds with the host cell surface Angiotensin-converting enzyme 2 (ACE2) facilitating virus entry, invading and replication.[1][5][6][7][8][9][10].Further analysis even suggested that COVID-19 recognizes human ACE2 more efficiently than SARS-CoV increasing the ability of COVID-19 to transmit from human to human [11][12] Upregulation of human ACE2 enhanced and induced disease severity in a mouse model of SARS-CoV infection, demonstrating that viral entry into cells is a critical step[13][14] Receiving Vaccine based on COVID-19 spike protein may increase the risk of Cellular ACE2 autoimmunity via production of autoantibodies . Many studies demonstrated that autoimmune response to Angiotensin-converting enzyme 2 ( ACE2) induced by forced presentation of the ACE2 protein in a complex with CoV Spike protein in Fc Receptor positive Antigen Presenting Cells in the lung [3][4] According to this we hypothesis that spike proteins produced by Vaccine based on the spike protein which would potentially bind to the elevated levels of soluble ACE2 enzyme. This complex of spike protein with multiple soluble ACE2 enzymes which is similar to COVID-19 binding with cellular and soluble ACE2 will be presented to macrophages to highlight antigens for antibody production. It is very possible that Abs will be produced that target the Angiotensin Converting Enzyme 2 of host cells enzyme. The combination of the virus spike protein or vaccine spike protein with the soluble ACE2 receptor becomes antigenic, which may cause the formation of antibodies against not only the virus spike protein or vaccine spike protein , but also parts of the ACE and ACE2 receptor. Therefore we hypothesize that Vaccines based on the spike protein might initiate Autoantibodies and T cells to ACE2 via binding of spike protein particles produced by vaccine with its receptors ACE2 and The development of autoantibodies to ACE2 might make damage to the host epithelial cell in lungs and the other different organs which express ACE2 in lung, heart and kidney would lead to inflammation at those sites. This pattern of lung injury also occurs in Pulmonary Hypertension secondary to Scleroderma with elevated levels of anti ACE2 antibodies.[73][78].In addition, we expect that any drug upregulation of ACE2 as in diabetic and hypertensive patients will increase the risk of autoantibodies in case of immunization by Vaccine based on the COVID-19 spike protein. As a result we think that covid-19 vaccine developer should use a suitable ACE2 modulator to decrease this possible risk via helping in formation of antibodies targeting spike protein not antibodies targeting ACE2 and spike protein complex which may increase the risk of cellular ACE2 auto antibodies , The COVID-19 vaccine may be altered each year to counter changes to circulating strains therefore, the possible risk of cellular ACE2 damage by autoantibodies produced by vaccine based on COVID-19 vaccine may increase with vaccination .After searching, we found a study analyzed a broad set of 672 clinically approved drugs for treatment in cell lines demonstrated that isotretinoin was the potent and strongest downregulator of Angiotensin-converting enzyme 2 (ACE2) receptors [15] and further, studies reported that it may prevent the cellular entry of SARS-CoV-2 and can be a taken as a targeted therapy in COVID-19 [16][17][18]. The primary isomers of RA formed in vivo are 9-cis-retinoic acid (9cRA) and All-trans-Retinoic Acid (atRA) and; each binds separate RA receptor types, thus acting upon a select subset of genes [76]. 13cRA is a synthetic form that may function similar to the other produced isoforms, or by isomerization to atRA and 9c RA. Although the exact mechanism of action is unclear; in other words, therefore we hypothesis that isotretinoin binds directly to ACE2 receptors and leads to its downregulation via blocking ACE2 binding capacity and this mechanism may lead to block of COVID-19 binding to cellular and soluble ace2 receptors

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18-40 years.
2. Increased risk of SARS-CoV-2 infection
3. Medically stable

Exclusion Criteria:

1. Confirmed or suspected immunosuppressive or immunodeficient state
2. Prior or concomitant vaccine therapy for COVID-19
3. significant disease, disorder, or finding
4. Hypercholesterolemia
5. Hypertriglyceridemia
6. Liver disease
7. Renal disease
8. Sjögren syndrome
9. Pregnancy
10. Lactation
11. Depressive disorder
12. Body mass index less than 18 points or higher than 25 points
13. Contraindications for hormonal contraception or intrauterine device.
14. Autoimmune diseases A history of organ, bone marrow or hematopoietic stem cell transplantation
15. Patients receiving anti-hcv treatment
16. Permanent blindness in one eye
17. History of iritis, endophthalmitis, scleral inflammation or retinitis 15-90 days of retinal detachment or eye surgery
18. The competent physician considered it inappropriate to participate in the study

    -------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------

Safety and promising features of isotretinoin in tne era of COVID 2019 according Principal Investigator Protocol:

1. This medication have the feature of Aerosolized Drug Delivery to increase its efficacy beside Oral administration, Which makes it distinct from other medication in which should dose be only given orally. A study demonstrated that treating with 13 cis retinoic acid aerosolized via inhalation rout did not cause any damage in lung cells.
2. Repeated high doses of 13 cis retinoic by inhalation resulted in moderate loss of body weight, but microscopic investigation of ten tissues including lung and oesophagus did not detect any significant aerosol-induced damage. The results suggest that administration of isotretinoin via powder aerosol inhalation is probably superior to its application via the oral route in terms of achieving efficacious drug concentrations in the lung.
3. Inhaled isotretinoin might provide sufficient drug to the target cells for efficacy while avoiding systemic toxicity.
4. A study demonstrated that 13 cis retinoic is used in treating Emphysema (emphysema is a lung condition that causes shortness of breath)
5. RA has been reported to induce formation of new alveoli and returns elastic recoil in the lung to approximately normal values in animal models of emphysema.
6. Strong expectation of complete COVID -19 blockade from cell entry and infection depending on strong ethics, researches and references.
7. Availability of our compounds.
8. Ease of application.
9. Expectation of COVID -19 treating by isotretinoin via more than one distinct mechanism.
10. Inhibiting of thrombosis and platelet which is the most serious consequences caused by viral spike protein or vaccine spike protein:- Co-incubation with 13-cis-RA and IL-1 resulted in a synergic increase in the release of Prostacyclin Synthase (PGI2). PGI is a powerful vasodilator that inhibits platelet aggregation through activation of adenylate cyclase,Consistently 13-cis-RA increased the ability of HUVEC to inhibit Arachidonic acid -induced platelet aggregation. Because of 13cRA is a synthetic form that may function similar to the other produced isoforms, or by isomerization to atRA and 9c RA. RA therapy has proven anti-platelet , anti- inflammatory, and fibrinolytic activities we suggest that 13cRA may protect patients infected with covid-19 from pulmonary clots.
11. Isotretinoin can induce Innate Immune response for recognition of CoV in addition to , inhibiting IL-6 The genome of Middle East Respiratory Syndrome Coronavirus is recognized by melanoma differentiation-associated protein-5 (MDA5), retinoic acid inducible gene-1 (RIG-1) and endosomal toll-like receptor 3 (TLR3) as pathogen-associated molecular patterns which recognize ssRNA and dsRNA intermediate of COVID-19.This recognition resulted in the formation of type-1 interferon (IFN1) as in (fig 6).COVID-19 synthesizes proteins that hinder the production IFN1 in its replication pathway, which is an evasion mechanism [123],[124],[125],[126],[127],[128],[129]. A study demonstrated that TLR3(-/-), TLR4(-/-), and TRAM(-/-) mice are more susceptible to SARS-CoV than wild-type mice but experience only transient weight loss with no mortality in response to infection. On the other hand, mice deficient in the TLR3/TLR4 adaptor TRIF are highly susceptible to SARS-CoV infection, showing increased weight loss, mortality, reduced lung function, increased lung pathology, and higher viral titers [130]. Previous studies revealed that the high level of IFN- α/β produced via the TLR3-IRF3/IRF7 pathway and IFN-β is the reason for inhibiting Dengue virus (DENV) replication [131]. 13-cis retinoic acid induced significant upregulation of toll-like receptor 3 (TLR3), mitochondrial antiviral-signaling protein (MAVS) and (RIG-I) and IFN regulatory factor 1 expression in a time-dependent [132].Furthermore, A study reported that 13-cis-retinoic acid and other retinoid analogs inhibit IL-1-induced IL-6 production and that this effect is analog-specific and, at least partially, transcriptionally mediated. This effect was dose-dependent with an IC50 of 10(-7) M RA and significant inhibition was found with doses of RA as low as 10(-8) M [122].

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy of the candidate oral and aerosolized isotretinoin for providing complete protection against COVID-19 in adults aged 18 years and older. | Time Frame: Study duration (12 months from last dose donation ) ]
  Occurrence of COVID-19 infection
Assess the safety of the candidate spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine in adults aged 18 years and older. | Time Frame: Study duration (24 months from last vaccination) ]
  Occurrence of expected serious side effects throughout the study duration and in the duration of followup:
  1. Generation of Autoantibodies against host ACE2
  2. Platelets aggregation
  3. Thrombosis
  4. Lung damage and fibrosis
  5. Sexual problems
  6. Neurological problems
Assess the efficacy of the candidate vaccine spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine for providing complete protection against COVID-19 in adults aged 18 years and older. | Time Frame: Study duration (12 months from last dose donation ) ]
  Occurrence of COVID-19 infection
Assess the efficacy of the candidate spike protein based vaccine such as ChAdOx1 nCoV-19 combined with oral and aerosolized isotetinoin in adults aged 18 years and older. for providing complete protection against COVID-19 | Time Frame: Study duration (12 months from last dose donation ) ]
  Occurrence of COVID-19 infection
Assess the safety of the candidate spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine in combination with oral or aersolized 13 cis retinoic acid in adults aged 18 years and older. | Time Frame: Study duration (24 months from last vaccination) ]
  Occurrence of expected serious side effects throughout the study duration and in the duration of followup:
  1. Generation of Autoantibodies against host ACE2
  2. Platelets aggregation
  3. Thrombosis
  4. Lung damage and fibrosis
  5. Sexual problems
  6. Neurological problems

SECONDARY OUTCOMES:
Assess efficacy of the candidate oral and aerosolized isotretinoin against COVID-19 | Time Frame: Study duration (12 months from last dose donation ) ]
  Number of intensive care unit (ICU) admissions associated with COVID-19
Assess efficacy of the candidate spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine against COVID-19 | Time Frame: Study duration (12 months from last dose donation ) ]
  Number of intensive care unit (ICU) admissions associated with COVID-19
Assess safety of the candidate spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine combined with oral and aerosolized isotetinoin in vaccinated participants | Time Frame: Study duration (48 months from last vaccination) ]
  Number of intensive care unit (ICU) admissions associated with COVID-19
Assessment the expression of MDAP-5 , RIG-1 , IFN1, TLR3 and IFN1 in Isotretinoin treated participants in comparison with vaccinated participants with spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine | Time Frame: Study duration (12 months from last dose donation ) ]
Absolute lymphocyte counts (CD4,CD8 and CD25+FOXP3+ Regulatory T cells ) in Isotretinoin treated participants in comparison with vaccinated participants with spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine | Time Frame: Study duration (12 months from last dose donation ) ]
Assessment the generated IgA antibodies in Isotretinoin treated participants in comparison with vaccinated participants with spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine | Time Frame: Study duration (12 months from last dose donation ) ]
Thrombin | Time Frame: Study duration (12 months from last dose donation ) ]
  Thrombin time (TT)
  Isotretinoin therapy has furthermore proven anti-inflammatory, anti-platelet and fibrinolytic activities. which may protect participants from widespread blood clots in case of infection with covid-19
Assessment the expression of Transe membrane protease ,serine II (TMPRSS2) changes over time in Isotretinoin treated participants in comparison with vaccinated participants with spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine | Time Frame: Study duration (12 months from last dose donation ) ]
Assessment the expression of Angiotensin-converting enzyme II (ACE2) changes over time in Isotretinoin treated participants in comparison with vaccinated participants with spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine | Time Frame: Study duration (12 months from last dose donation ) ]
Platelet aggregation in Isotretinoin treated participants in comparison with vaccinated participants with spike protein based vaccine such as ChAdOx1 nCoV-19 vaccine | Time Frame: Study duration (24 months from last vaccination) ]
ACE2 autoantibodies IgG and IgM | Time Frame: Study duration (24 months from last vaccination) ]

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Elkazzaz, M.Sc in Biochemistry, Principal Investigator — Facculty of Science, Damietta University